CLINICAL TRIAL: NCT01566071
Title: Ability to Drive of Early Stage Alzheimer Disease
Acronym: DRIVE COG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: PN11009
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2016-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Assessment of drive abilities

SUMMARY:
The main objectives of this study are:

* To evaluate the driving capacities in a population of elderly subjects with early stage Alzheimer Disease (AD) in a real-life situation.
* Define a typology of the main errors made in this population.
* Propose adaptive measures or technological aids that would make it possible for these patients to maintain their ability to drive a car while limiting risk.

ELIGIBILITY:
Inclusion Criteria:

The following subjects will be included and classified as " patients " :

* Age > 70 years
* With established diagnosis of Alzheimer's disease as defined by DSM IV
* With MMSE score ≥ 24 (early-stage Alzheimer's disease)
* Holder of a valid driving license
* With regular driving activity (drives at least once per week)
* Informed consent provided.

The following subjects will be included and classified as " controls " :

* Age > 70 years,
* Absence of cognitive impaired that interferes with their daily life at initial evaluation,
* Holder of a valid driving license,
* With regular driving activity (drives at least once per week),
* Informed consent provided.

Exclusion Criteria:

* Dementia syndrome(s) other than Alzheimer's disease,
* MMSE score < 24
* Informed consent not provide

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JEAN-LUC NOVELLA, MD PhD, Principal Investigator — CHU de Reims
Locations (1):
- CHU de REIMS, Reims, France, France

REFERENCES:
- [Background] Paire-Ficout L, Lafont S, Conte F, Coquillat A, Fabrigoule C, Ankri J, Blanc F, Gabel C, Novella JL, Morrone I, Mahmoudi R. Naturalistic Driving Study Investigating Self-Regulation Behavior in Early Alzheimer's Disease: A Pilot Study. J Alzheimers Dis. 2018;63(4):1499-1508. doi: 10.3233/JAD-171031. PMID 29782312